CLINICAL TRIAL: NCT01686581
Title: A 24-month, Prospective, Non-interventional Study to Describe the Long Term, Real-Life Use of BOTOX® for the Symptomatic Treatment of Adults With Chronic Migraine, Measuring Healthcare Resource Utilization, and Patient Reported Outcomes Observed in Practice
Brief Title: An Observational Study of BOTOX® as Headache Prophylaxis for Chronic Migraine
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: MAF/AGN/NS/CM/002
Record Dates: First submitted 2012-09-13; First posted 2012-09-18 (Estimated); Results first posted 2018-11-09 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-04

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BOTOX®: BOTOX® (botulinum toxin Type A) administered according to physician prescription for the treatment of chronic migraine; all treatment decisions lie with the physician.
  Interventions: Drug: botulinum toxin Type A

INTERVENTIONS:
Drug: botulinum toxin Type A — Botulinum toxin Type A (BOTOX®) administered according to physician prescription.
  Other Names: BOTOX®; onabotulinumtoxin A

SUMMARY:
This is an observational study to describe the long term use of Onabotulinumtoxin A (BOTOX®) as prescribed by the physician for headache prophylaxis in adults with chronic migraine. All treatment decisions lie with the physician.

ELIGIBILITY:
Inclusion Criteria:

- Prescribed BOTOX® for the prophylaxis of headaches.

Exclusion Criteria:

* Received treatment with any botulinum toxin Type A serotype in the last 26 weeks
* Current participation in Allergan's Botox Chronic Migraine Post-Authorisation Safety Study (protocol 191622-110).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic migraine prescribed BOTOX® for the prophylaxis of headaches
Sampling Method: Non-Probability Sample
Enrollment: 641 (Actual)
Dates: Start 2012-07-23 (Actual); Primary Completion 2016-10-12 (Actual); Study Completion 2016-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (77):
- Germany (56):
  - Nicole Strickling, Aachen
  - Manfred Oberling, Bad Camberg
  - Kathrin Krome, Bamberg
  - Heike Förster, Baunatal
  - MVZ Schmerzzentrum Berlin, Berlin
  - Christoph Engelmann, Berlin
  - Andreas Kupsch, Berlin
  - Hans-Dieter Zug, Böblingen
  - Andreas Schwittay, Böhlen
  - Bezirksklinikum Mainkofen, Deggendorf
  - Ulrike Kirchhöfer, Erfurt
  - Michael Kiszka, Erfurt
  - Astrid Gendolla, Essen
  - Jürgen Hamacher, Essen
  - Schmerzzentrum Rhein Main in Frankfurt, Frankfurt
  - Bernhard Hellwig, Freiburg im Breisgau
  - G. Müller-Schwefe, Göppingen
  - Borries Kukowski, Göttingen
  - Peter Asmus, Guelders
  - Veit Becker, Hamburg
  - Hanno Jaeger, Hamburg
  - Klaus Gerlach, Hanover
  - Medizinische Hochschule Hannover, Hanover
  - Ulrike Köhler, Heidelberg
  - Frank Halbgewachs, Heidenheim
  - Dirk Buschmann, Herford
  - Rotes Kreuz Krankenhaus Kassel, Kassel
  - Schmerzklinik Kiel, Kiel
  - Migräne-Klinik Königstein, Königstein
  - Neuroscience Center Leipzig, Leipzig
  - Dietmar Walter Noack, Limburgerhof
  - Lothar Klimpel, Limburgerhof
  - St.-Marien-Hospital GmbH, Lünen
  - Olaf Günther, Magdeburg
  - Institut für Forschung und Prävention, Mainz
  - Stephan Nautscher-Timmermann, Mühlhausen
  - Praxis für Neurologie und SchmerzMedizin, München
  - Matthias Haslbeck, München
  - Klinikum der Universität München - Großhadern, Neurologische Klinik, München
  - Neurologie und Kopfschmerzzentrum Münchner Freiheit, München
  - Schmerztherapiezentrum Münster, Münster
  - Roland Leger, Nuremberg
  - Dr. Becker Rhein-Sieg-Klinik, Nümbrecht
  - Matthias Röder, Oberhausen
  - mediPlan Klinik GmbH, Ostfildern
  - Frank Freitag, Potsdam
  - Universität Rostock, Klinik für Neurologie, Rostock
  - Ingo Palutke, Stadtroda
  - Heinz Peter Herbst, Stuttgart
  - Anselm Kornhuber, Ulm
  - Universitätsklinikum Ulm, Klinik für Neurologie, Ulm
  - Volker Heinicke, Weimar
  - Parkinson-Klinik Wolfach, Wolfach
  - Michaela Krause, Wolfratshausen
  - Jochen Ulzheimer, Würzburg
  - Dorothea Händel, Zwickau
- Italy (3):
  - Ospedale Careggi, Florence
  - Istituto Neurologico Carlo Besta di Milano, Milan
  - Azienda Ospedaliera Sant'Andrea, Roma
- Hodeverket Headache Clinic, Sandnes, Norway
- Russia (5):
  - LLC Neyroklinika, Khabarovsk
  - LLC Center for Interdisciplinary Dentistry and Neurology, Moscow
  - LLC Clinic Sesil +, Moscow
  - LLC University Headache Clinic, Moscow
  - LLC Sibneuromed, Novosibirsk
- Spain (6):
  - Hospital Universitario de Burgos, Burgos
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Central de Asturias, Oviedo
  - Hospital Santiago de Compostela, Santiago de Compostela
  - Hospital Galdácano, Usansolo
- Sweden (3):
  - Löfvingkliniken, Gothenburg
  - Centralsjukhuset i Karlstad, Karlstad
  - Läkarhuset Utsikten, Stockholm
- United Kingdom (3):
  - Spire Hull and East Riding Hospital, Anlaby
  - University Hospital of North Staffordshire, Neurology Research Unit, Stoke-on-Trent
  - Mid Yorkshire NHS Trust, Wakefield

REFERENCES:
- [Derived] Ahmed F, Gaul C, Kollewe K, Singh RC, Sommer K. Real-World Safety and Efficacy of 156 U - 195 U OnabotulinumtoxinA in Adults With Chronic Migraine: Results From the REPOSE Study. BMC Neurol. 2025 May 6;25(1):197. doi: 10.1186/s12883-025-04087-7. PMID 40329224
- [Derived] Kollewe K, Gaul C, Gendolla A, Sommer K. Real-life use of onabotulinumtoxinA reduces healthcare resource utilization in individuals with chronic migraine: the REPOSE study. J Headache Pain. 2021 Jun 2;22(1):50. doi: 10.1186/s10194-021-01260-4. PMID 34078259
- [Derived] Ahmed F, Gaul C, Garcia-Monco JC, Sommer K, Martelletti P; REPOSE Principal Investigators. An open-label prospective study of the real-life use of onabotulinumtoxinA for the treatment of chronic migraine: the REPOSE study. J Headache Pain. 2019 Mar 7;20(1):26. doi: 10.1186/s10194-019-0976-1. PMID 30845917

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BOTOX®
Started | 641
Safety Analysis Set; Received Study Drug | 633
Completed 24 Months | 128
Completed (Completed=Completed Treatment) | 464
Not Completed | 177
Not completed — Side-effects or Health Problems | 15
Not completed — Lack of Efficacy | 90
Not completed — Participant Concerned about Risks | 6
Not completed — Thinks Injections Too Painful | 8
Not completed — Thinks Injections Take Too Much Time | 2
Not completed — Trying to get Pregnant or Nursing | 2
Not completed — Thinks it is Inconvenient | 17
Not completed — Other Miscellaneous Reasons | 36
Not completed — Reason Missing | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who received at least one dose of BOTOX®.
Arm/Group | BOTOX®
Number analyzed (Participants) | 633
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 540
  Male | 93

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Admitted to the Hospital for Headache
Description: The Baseline value included participants who had been admitted to the hospital for headache in the last 3 months prior to the baseline visit (first administration of BOTOX®); the Last Follow-up value included participants who been admitted to the hospital for headache since the previous visit.
Time Frame: Baseline (previous 3 months prior to first dose of BOTOX®) and Last Follow-up Visit (FU last) [median 21.20 months]
Population: Participants from the Safety Analysis Set, all participants who received at least one dose of BOTOX®, with data available for analysis at the given time-point.
Measure: Number; unit: percentage of participants
Arm/Group | BOTOX®
Number analyzed (Participants) | 633
percentage of participants
  Baseline | 6.0
  FU last: number analyzed (Participants) | 607
  FU last | 2.1

2. Primary Outcome: Mean Number of Days of Headache-related Hospital Admissions
Description: The number of admission days is presented as the mean, normalized to a period of 90 days. The Baseline value included admissions during the last 3 months prior to the baseline visit (first administration of BOTOX®); the Last Follow-up value included admissions since the second-to-last visit.
Time Frame: Baseline (previous 3 months prior to first dose of BOTOX@) to FU last [median 21.20 months]
Population: Participants from the Safety Analysis Set, all participants who received at least one dose of BOTOX®, who were hospitalized.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | BOTOX®
Number analyzed (Participants) | 38
days
  Baseline | 8.9 (20.14)
  FU last: number analyzed (Participants) | 13
  FU last | 4.8 (10.98)

3. Primary Outcome: Percentage of Participants Who Visited Any Healthcare Professional (HCP)
Description: The Baseline value included participants who had visited an HCP in the last 3 months prior to the baseline visit (first administration of Botox); the value for FU last included participants who visited an HCP since the second-to-last visit.
Time Frame: Baseline (previous 3 months prior to first dose of BOTOX®) to FU last [median 21.20 months]
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | BOTOX®
Number analyzed (Participants) | 633
percentage of participants
  Any HCP Visit: Baseline | 45.8
  Any HCP Visit: FU last: number analyzed (Participants) | 607
  Any HCP Visit: FU last | 17.1
  Primary Care Consultant Visit: Baseline | 30.6
  Primary Care Consultant Visit: FU last: number analyzed (Participants) | 607
  Primary Care Consultant Visit: FU last | 12.7
  Outpatient Consultation: Baseline | 33.3
  Outpatient Consultation: FU last: number analyzed (Participants) | 607
  Outpatient Consultation: FU last | 6.8
  Accident and Emergency Visit: Baseline | 6.3
  Accident and Emergency Visit: FU last: number analyzed (Participants) | 607
  Accident and Emergency Visit: FU last | 2.6
  Alternative Practitioner: Baseline | 6.3
  Alternative Practitioner: FU last: number analyzed (Participants) | 607
  Alternative Practitioner: FU last | 2.0
  Other: Baseline | 4.3
  Other: FU last: number analyzed (Participants) | 607
  Other: FU last | 0.5

4. Secondary Outcome: Change From Baseline in Migraine-Specific Quality of Life Questionnaire (MSQ) Score
Description: The MSQ is a 14-item questionnaire to measure health-related quality-of-life attributed to migraine in the past 4 weeks. Each item is scored on a 6-point scale where: 1=none of the time to 6=all of the time. There are 3 dimensions: Role-function Restrictive (questions 1 to 7; score range 7 to 42), Role-function Preventive (questions 8 to 11; score range 4 to 24) and Emotional-function (questions 12 to 14; score range 3 to 18). The individual dimension scores were converted to a score of 0 to 100; the total score ranged from 0 to 300 with higher numbers representing a better quality of life. A positive change from baseline in the dimension scores and the total score indicates that quality of life has improved.
Time Frame: Baseline to Last Administration of BOTOX® (ADM last) [median 20.30 months]
Population: Safety Analysis Set, all participants who received at least one dose of BOTOX®, with data available for analysis at the given time-point.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | BOTOX®
Number analyzed (Participants) | 633
score on a scale
  Role Function-Restrictive: Baseline (BL): number analyzed (Participants) | 591
  Role Function-Restrictive: Baseline (BL) | 37.14 [0.0 to 100.0]
  Role Function-Restrictive: Change BL to ADM last: number analyzed (Participants) | 537
  Role Function-Restrictive: Change BL to ADM last | 25.71 [-28.6 to 97.1]
  Role Function-Preventive: Baseline: number analyzed (Participants) | 586
  Role Function-Preventive: Baseline | 50.0 [0.0 to 100.0]
  Role Function-Preventive: Change BL to ADM last: number analyzed (Participants) | 550
  Role Function-Preventive: Change BL to ADM last | 20.00 [-55.0 to 100.0]
  Emotional Function: Baseline: number analyzed (Participants) | 593
  Emotional Function: Baseline | 40.00 [0.0 to 100.0]
  Emotional Function: Change from BL to ADM last: number analyzed (Participants) | 552
  Emotional Function: Change from BL to ADM last | 26.67 [-60.0 to 100.0]
  Total Score: Baseline: number analyzed (Participants) | 583
  Total Score: Baseline | 132.86 [0.0 to 300.0]
  Total Score: Change from BL to ADM last: number analyzed (Participants) | 529
  Total Score: Change from BL to ADM last | 70.95 [-96.2 to 297.1]

5. Secondary Outcome: Change From Baseline in the EQ-5D Questionnaire Total Score
Description: The EQ-5D consists of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) assessed by the participant using a 3-point scale: 1=no problems, 2=some problems and 3=extreme problems. The combination of levels from the 5 dimensions results in a health state code. The total score is calculated by converting the health state code into a score: start with score 1.000=[11111] (perfect health state), subtract 0.081 (constant) for any other state, subtract nothing for level 1 on any dimension, subtract appropriate level 2 or level 3 value for each dimension from a table of constants [Level 2: Mobility 0.069, Self-care 0.104, Usual activity 0.036, Pain/discomfort 0.123, Anxiety/depression 0.071] [Level 3: Mobility 0.314, Self-care 0.214, Usual activity 0.094, Pain/discomfort 0.386, Anxiety/depression 0.236], subtract 0.269 if any dimension has a level 3 problem. Higher numbers indicate better health. A positive change from Baseline indicates improvement.
Time Frame: Baseline (prior to first dose of BOTOX®) to ADM last [median 20.30 months]
Population: Participant from the Safety Analysis Set, all participants who received at least one dose of BOTOX®, with data available at the given time-point.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | BOTOX®
Number analyzed (Participants) | 633
score on a scale
  Baseline: number analyzed (Participants) | 596
  Baseline | 0.69 [-0.59 to 1.0]
  Change from Baseline to ADM last: number analyzed (Participants) | 531
  Change from Baseline to ADM last | 0.107 [-0.889 to 1.390]

6. Secondary Outcome: Change From Baseline in the Health State Score of the EQ-5D Questionnaire
Description: The EQ-5D health state scale is a visual analog scale that ranges from 0 (worst imaginable health state) to 100 (best imaginable health state), with higher scores indicating a better state of health. Participants were asked to rate their health state on a drawn line that started at 0 and ended at 100. A positive change from baseline in the health state score indicates that the participant's health state has improved.
Time Frame: Baseline (prior to first dose of BOTOX®) to ADM last [median 20.30 months]
Population: Participants from the Safety Analysis Set, all participants who received at least one dose of BOTOX®, with data available at the given time-point.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | BOTOX®
Number analyzed (Participants) | 633
score on a scale
  Baseline: number analyzed (Participants) | 582
  Baseline | 50.0 [0 to 100]
  Change from Baseline to ADM last: number analyzed (Participants) | 519
  Change from Baseline to ADM last | 10.0 [-86 to 91]

7. Secondary Outcome: Change From Baseline in the Number of Headache Days
Description: At each visit, participants were asked to provide the number of headache days he/she experienced in the last month. A headache day was defined as 4 or more hours of continuous headache. A negative change from Baseline (less headache days) indicates improvement.
Time Frame: Baseline (prior to first dose of BOTOX®) to ADM last [median 20.30 months]
Population: as for outcome 6
Measure: Median (Full Range); unit: days
Arm/Group | BOTOX®
Number analyzed (Participants) | 633
days
  Baseline | 20.0 [8 to 31]
  Change from Baseline to ADM last: number analyzed (Participants) | 571
  Change from Baseline to ADM last | -11.0 [-30 to 15]

8. Secondary Outcome: Percentage of Participants With Good or Very Good Responses on the 4-Point Treatment Satisfaction Scale
Description: At each visit, participants and physicians were asked to indicate the level of satisfaction that he/she had with the treatment. Physicians indicated the level of satisfaction with the patient's treatment. The 4- point scale consisted of the following responses: insufficient, moderate, good and very good. The combined percentage of "good" and "very good" responses by participants and physicians are reported.
Time Frame: ADM last [median 20.30 months]
Population: Participants from the Safety Analysis Set, all participants who received at least one dose of BOTOX®, with data available.
Measure: Number; unit: percentage of participants
Arm/Group | BOTOX®
Number analyzed (Participants) | 571
percentage of participants
  Physician Assessment | 78.1
  Patient Assessment | 76.0

ADVERSE EVENTS:
Time Frame: First dose of study drug to FU last [median 21.20 months]
Description: As per the protocol, Adverse Drug Reactions and Serious Adverse Drug Reactions were collected.
Arm/Group | BOTOX®
All-Cause Mortality (participants affected / at risk) | 0/633
Serious Adverse Events (participants affected / at risk) | 8/633
Other Adverse Events (participants affected / at risk) | 34/633
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BOTOX® (N=633)
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1
Mental disorder (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1
Psychosomatic disease (Psychiatric disorders) | 1
Migraine (Nervous system disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Headache (Nervous system disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BOTOX® (N=633)
Eyelid ptosis (Eye disorders) | 34

LIMITATIONS AND CAVEATS:
There were no Primary or Secondary Outcome Measures specified in the protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.